CLINICAL TRIAL: NCT03442816
Title: Evaluation of a Metabolic Hyperspectral Retinal Camera (MHRC) in Spectrally Resolved Reflectance and Fluorescence Imaging in a Diverse Population
Brief Title: Retinal Metabolic Imaging in a Diverse Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor no longer supported this study
Sponsor: Optina Diagnostics Inc. (Industry)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 050317
Record Dates: First submitted 2018-02-13; First posted 2018-02-22 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2019-09

CONDITIONS: Technical Capabilities of the Device

STUDY DESIGN:
Intervention Model Description: Subjects will undergo 1) an ophthalmic evaluation and 2) an evaluation with the device (camera)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MHRC camera (Experimental): Subjects will undergo a retina imaging session with the MHRC camera.
  Interventions: Device: MHRC Camera

INTERVENTIONS:
Device: MHRC Camera — Evaluate the technical capabilities of the device to obtain quality images in reflectance and fluorescence imaging modes in a diverse population.

SUMMARY:
This research project aims to evaluate use in a clinical context of a novel imaging instrument, the Metabolic Hyperspectral retina Camera (MHRC) from Optina Diagnostics. This camera enables the acquisition of retinal images at multiple colors (up to 100 specific colors) and therefore extract way more information that can be captured with a conventional retinal camera (up to 3 colors). This additional color information available for each pixel of the image could be useful to identify signs of pathologies having manifestations in the retina. The performances of this new prototype camera will be evaluated and the acquisition procedures optimized in a diverse population of subjects.

DETAILED DESCRIPTION:
Hyperspectral retinal imaging results from several consecutive images taken while the filter scans a wide spectral range to obtain one spectrum for each image pixel. The combination of imaging and spectroscopy offered by hyperspectral imaging makes it possible to identify and quantify several specific biomolecules in the retina and the optic nerve, thus paving the way for metabolic imaging of the fundus. Subsequent analysis of the light signal with algorithms and image analysis software tools permits extracting molecular information modulated according to the underlying pathology. This technique thus permits direct, non-invasive and inexpensive diagnosis of pathologies of the retina and systemic pathologies presenting manifestations in the eye.

In this research project, Optina Diagnostics aims to evaluate in a clinical context a novel Metabolic Hyperspectral Retinal Camera (MHRC) based on a mydriatic camera customized for observation of the fundus in combination with a tunable filter, i.e., one permitting selection of a specific wavelength, in order to provide monochromatic light in the visible and near infrared spectrum (energy spectrum between 450 and 900 nm).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and up with vision in at least one eye.

Exclusion Criteria:

* Inadequate pupil dilation (< 6mm diameter) or contraindicated
* Deficient visual fixation
* Refractive error outside the -9 to +9 range
* Media opacities or intraocular bleeding preventing retinal imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2020-09-26 (Actual)

PRIMARY OUTCOMES:
Quality images in reflectance and fluorescence | 1 day visit
  Evaluate the technical capabilities of the device to obtain quality images in reflectance and fluorescence imaging modes in a diverse population .

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kertes, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No